CLINICAL TRIAL: NCT01008163
Title: A Phase Ⅱ, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding, Efficacy and Safety of YY-351 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Dose-Finding, Efficacy and Safety Study of YY-351 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuyu Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YY351-1; YY-351-4
Record Dates: First submitted 2008-10-20; First posted 2009-11-04 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): YY-351, PO, 1T tid. / Placebo, 1T tid.
  Interventions: Drug: YY-351/Placebo
- 2 (Experimental): YY-351. PO, 2T bid. / Placebo 2T qd.
  Interventions: Drug: YY-351/Placebo
- 3 (Experimental): YY-351, PO, 2T tid.
  Interventions: Drug: YY-351
- 4 (Placebo Comparator): Placebo, PO, 2T tid.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YY-351/Placebo — comparison of different dosages of drug
  Other Names: Ginsam
  Arms: 1
Drug: YY-351/Placebo — comparison of different dosages of drug
  Other Names: Ginsam
  Arms: 2
Drug: YY-351 — comparison of different dosages of drug
  Other Names: Ginsam
  Arms: 3
Drug: Placebo — comparison of different dosages of drug
  Arms: 4

SUMMARY:
The purpose of this trial is to determine the dosage selected and to evaluate the efficacy and safety of YY-351.

DETAILED DESCRIPTION:
Ginseng has been widely studied for treatment of diabetes, dyslipidemia and obesity. Interestingly, in addition to ginseng root, ginseng berry and leaf were also shown to reduce blood glucose in diabetic models. In our recent study, ginsam, vinegar extraction from Panax ginseng, which is enriched in the ginsenoside Rg3, has distinct beneficial effects on glucose metabolism and body weight control in an obese animal model of insulin resistance by changing the expression of genes involved in glucose and fatty acid metabolism. Our group has also published that Rg3 improves insulin signaling and glucose uptake primarily by stimulating the expression of IRS-1 and GLUT4. Thus, we have evaluated the efficacy, dose-response relationships and safety of a ginsam, a vinegar extract from Panax ginseng.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of Type 2 diabetes(more than 3months)
* Patients aged over 18 years
* FPG levels in the range : 126 - 270mg/dL or HbA1c : 7.0 - 12.0%

Exclusion Criteria:

* Pregnant women, Breast feeding, or actively trying to be come pregnant
* Patients with Type 1 DM, gestational diabetes or secondary diabetes
* FPG levels in the range : ≥ 270mg/dL HbA1c : < 7.0, >12.0%
* Patient who take the medicine which may affect to blood sugar control (i.e.systemic glucocorticoid)
* Patients with diabetic complications or the history of a case that would affect to efficacy and safety evaluation (i.e. Thyroid disorder, Cushing's Syndrome, Multiple ovarian cystoma, pheochromocytoma)
* Patients with Chronic hepatitis, hepatitis B, C (except healthy HBV carrier) or Liver diseases (AST or/and ALT >2 × ULN(upper limit normal))
* Patients with Kidney disorder (Cr>2.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the fasting plasma glucose and postprandial glucose [after 2 hours, oral glucose tolerance test (OGTT) (75 g)] and HbA1c | from baseline to Week 8

SECONDARY OUTCOMES:
Subjects achieving a glycemic response defined as ≤ 7.0% | from baseline to Week 8
Decrease of HbA1c > 0.5% | from baseline to Week 8
Biomarkers [liver function tests (LFT), high-sensitivity C-reactive protein (hsCRP), adiponectin] | from baseline to Week 8
Body weight (or body composition) | from baseline to Week 8
Waist girth | from baseline to Week 8
Homeostasis model assessment (HOMA) | from baseline to Week 8
Lipid profile | from baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD,PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Bungdang-Gu, South Korea